CLINICAL TRIAL: NCT00247039
Title: A Controlled Study to Determine The Clinical Efficacy Of Garlic Compounds In Patients With Chemotherapy Related Febrile Neutropenia
Brief Title: Garlic in Patients With Febrile Neutropenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moshe Gatt, Dr. Moshe Gatt, Hadassah Medical Organization
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 384 gar 1- HMO-CTIL; GAR1 (Other Grant/Funding Number: Dunsky grant for cancer research)
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Chemotherapy; Neutropenia
Keywords: neutropenia; fever; garlic; infection
MeSH Terms: conditions — Neutropenia; Fever; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Garlic extract (Experimental): Garlic extract capsules
  Interventions: Dietary Supplement: Solgar Israel
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Solgar Israel — Dietary Supplement: garlic natural compound one pill, 450 mg active garlic extract (Solgar, Israel), bid.
  Arms: Garlic extract
Other: Placebo capsules — placebo capsules
  Arms: Placebo

SUMMARY:
To determine the clinical effects of garlic in preventing and treatment of patients with chemotherapy related febrile neutropenia.These patients have a very high incidence of infections which are not routinely covered by the standard empiric therapy. Adding a non- toxic and possibly effective therapy may reduce the risk for infections, synergize the empiric antibiotic treatment and may lessen the need for broader spectrum and more severe side effects.

DETAILED DESCRIPTION:
Patients eligible are randomized to receive placebo or garlic capsules after chemotherapy course and until leukocyte recovery.

ELIGIBILITY:
Inclusion Criteria:

FN patients expected to have at least 5 days or more of neutropenia will be eligible for treatment with garlic compounds AST/ALT ≤ 3 times the upper limit of institutional laboratory normal.

Total bilirubin ≤ 2 times the upper limit of institutional laboratory normal.

BUN and creatinine should be ≤ 3 times the upper limit of institutional laboratory normal.

Newly diagnosed as well as previously treated patients will be eligible.

Exclusion Criteria:

History of clinically significant liver or kidney disease.

Patients on anti-coagulation therapy with Coumadin will be excluded because of the potential garlic interference with metabolism.

Patients receiving concomitant chemotherapeutic treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Time to fever and beginning of empiric antibiotic treatment. | 0-45 days post chemotherapy

SECONDARY OUTCOMES:
Documented and culture positive infections. | as above
Kind of infectious organisms and sensitivity to medicines. | as above
Length of infection | as above
Use of growth factors. | as above

CONTACTS AND LOCATIONS:
Overall Officials: moshe e gatt, dr, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Gatt ME, Strahilevitz J, Sharon N, Lavie D, Goldschmidt N, Kalish Y, Gural A, Paltiel OB. A Randomized Controlled Study to Determine the Efficacy of Garlic Compounds in Patients With Hematological Malignancies at Risk for Chemotherapy-Related Febrile Neutropenia. Integr Cancer Ther. 2015 Sep;14(5):428-35. doi: 10.1177/1534735415588928. Epub 2015 Jun 2. PMID 26036623